CLINICAL TRIAL: NCT05221216
Title: Single-center Retrospective Observational Study of Cotrimoxazole Dosing in Intensive Care Unit
Brief Title: Retrospective Observational Study of Cotrimoxazole Dosing in Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1452021/CHUSTE
Record Dates: First submitted 2021-12-31; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Acute Kidney Injury
Keywords: cotrimoxazole; Acute Kidney Injury; renal replacement therapy; pharmacodynamic
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients in Intensive Care unit: patients in Intensive Care unit with infection treated with cotrimoxazole will be included. Data will be collected of medical record.
  Interventions: Other: Collect data of medical record

INTERVENTIONS:
Other: Collect data of medical record — Collect data of medical record: plasma concentrations of cotrimoxazole, demographic data (age, weight, height), data on the use of an extra renal replacement therapy (RRT) (date, type, number of sessions and duration of extra renal replacement therapy (RRT))

SUMMARY:
Trimethoprim/sulfamethoxazole (TMP/SMX, cotrimoxazole) is the first-line therapy for Pneumocystis jirovecii pneumonia and bacterial infections in critically ill patients, where acute kidney injury (AKI) and renal replacement therapy (RRT) are regularly observed. Both may change half-life and subsequent concentrations. Specifically, Trimethoprim (TMP) is eliminated renally, whereas sulfamethoxazole (SMX) elimination is 80%metabolic/20%renal. Despite decades of cotrimoxazole use, data in acute kidney injury (AKI) are scarce and no consensus on dosing strategy has been established. Besides, pharmacodynamic parameter has not been determined, leading to an uncertainty on the dosing regimen.

DETAILED DESCRIPTION:
The objective is to compare the plasma concentrations of patients with acute renal failure (ARF) or requiring extra renal replacement therapy (RRT) with those of patients without these characteristics to look for differences in concentration.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in Intensive Care Units between October 2020 and July 2021 with infection treated with cotrimoxazole

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in Intensive Care Units between October 2020 and July 2021 with infection treated with cotrimoxazole will be included.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
plasma concentrations of cotrimoxazole (mg/l) | From the antibiotic initiation until the patient is discharged from the ICU with a maximal time frame of 10 weeks
  pharmacokinetic cotrimoxazole

CONTACTS AND LOCATIONS:
Overall Officials: Sophie PERINEL RAGEY, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No